CLINICAL TRIAL: NCT02528136
Title: The Clinical Carbetocin Myocardium Trial
Acronym: CMT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Leiv Arne Rosseland, Head for R&D department, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CarbeteocinHeart2014
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Pregnancy
MeSH Terms: interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbetocin (Experimental): One minute injection of carbetocin 100 µg after the delivery of the baby
  Interventions: Drug: Carbetocin
- Oxytocin (Active Comparator): One minute injection of oxytocin 2.5 U after the delivery of the baby
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Carbetocin
  Other Names: Pabal
  Arms: Carbetocin
Drug: Oxytocin
  Other Names: Syntocinon
  Arms: Oxytocin

SUMMARY:
Randomized comparison of different cardiotoxicity of carbetocin and oxytocin.

DETAILED DESCRIPTION:
Carbetocin has been in clinical use in EU for some years and the efficacy is documented in several RCTs. Circulatory adverse events leading to death has been reported after intravenous injection of oxytocin. Some studies indicate that oxytocin may lead to dose dependent ischemic ECG changes, prolongation of QT time and liberation of biomarkers of myocardial cell death. Previously we have demonstrated comparable vasodilatory effects of oxytocin and carbetocin. There is no clinical study comparing the specific myocardial effects of oxytocin with carbetocin. It may have great impact on the choice of standard medication if the cardiotoxicity of carbetocin is lower compared with oxytocin. The study of potential cardiotoxicity has to be performed in healthy women. Knowing that millions of laboring women have had uneventful injections of oxytocin and carbetocin after delivery, there is probably no reason to fear long lasting negative effects of either drug. If there are differences in cardiotoxicity, this new information should be taken into consideration when planning delivery in pregnant women with heart disease.

The aims of this study are to compare 0h (before C-section), 4h, 12h, 24h, and 48h plasma concentrations of Troponin I, Troponin T, proBNP, CK, and other relevant myocardial markers in elective healthy C-section patients randomized to oxytocin 2.5 U or carbetocin 100 µg, 1 minute injection immediately after delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy pregnant women age 18 to 50
2. Singleton pregnancy at gestational age 36 weeks or more
3. Able to read and understand Norwegian.

Exclusion Criteria:

1. Patients with placenta pathology such as praevia, acreta, pre-eclampsia
2. Patients with bleeding disorders including vonWillebrand disease type I.
3. Known intolerance to one of the two drugs.
4. Patients with prolonged QT-time or other serious cardiac diseases.
5. Liver or kidney failure.
6. Epilepsy.
7. Any medical reason why, in the opinion of the investigator, the patient should not participate

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
P-Troponin I | 48 hours
  P-Troponin I group differences

SECONDARY OUTCOMES:
P-Biomarkers | 48 hours
  P-Biomarkers group differences
ECG-changes | 1 hour
  Group differences in ECG-changes
Blood loss | 48 hours
  Calculated estimated blood loss (group differences in Hb change)

OTHER OUTCOMES:
Adverse events | 48 hours
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Pain intensity | 48 hours
  Group differences in pain intensity (Numeric rating scale 0 - 10) and consumption of PCA Morphine

CONTACTS AND LOCATIONS:
Overall Officials: Leiv Arne Rosseland, PhD, Study Director — Dep of Research and Development, Division of Emergencies and Critical Care, Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Division of Emergencies and Critical Care, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Participant data will be analyzed in the Research Group only

REFERENCES:
- [Derived] Bekkenes ME, Fagerland MW, Solberg OG, Aaberge L, Klingenberg O, Norseth J, Rosseland LA. Exploring cardiac effects after oxytocin 2.5 IU or carbetocin 100 mug: A randomised controlled trial in women undergoing planned caesarean delivery. Eur J Anaesthesiol. 2022 Dec 1;39(12):928-938. doi: 10.1097/EJA.0000000000001763. Epub 2022 Oct 17. PMID 36239406

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT02528136/Prot_SAP_000.pdf